CLINICAL TRIAL: NCT04851301
Title: Neural Mechanisms of Immersive Virtual Reality in Chronic Pain
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Luana Colloca, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00095888
Record Dates: First submitted 2021-04-06; First posted 2021-04-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pain; Virtual Reality; Placebo; Temporomandibular Disorder
Keywords: Naloxone; Observation; TMD volunteers; VR
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders | interventions — Exergaming; Naloxone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: AIM 1: This is a double-blinded, randomized, between- and within-subjects design (3 X 3) with TMD participants randomly assigned to one of three groups. The three groups are 1. Naloxone group 2. Saline group 3. Natural history group, in which participants will not be given any drugs. Within-subjects factor: All three groups will go through the following 3 conditions:1. Active VR (theBlu); 2. Sham VR; 3. No-VR.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The UM Pharmacy will assign de-identified study IDs to participants and provide the study drug (Naloxone or Saline) so that participants, the person conducting the experiment, and the investigator will be blind to the participant's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Naloxone (Active Comparator): NARCAN® Naloxone Nasal Spray will be used to determine how the opioid tone shapes VR-induced hypoalgesia. Participants will be stratified for sex and then randomized to naloxone (The dose of naloxone will be 4 mg, so 0.1 mL of 40 mg/ml naloxone solution given intranasally) or saline (0.1 mL 0.9% sodium chloride intranasally), respectively. Investigators, staff, and participants will be blinded to the treatment options.
  Interventions: Behavioral: Active Virtual Reality; Behavioral: sham Virtual Reality; Other: No Intervention; Drug: Naloxone
- Saline (Sham Comparator): Saline group, where participants will be given saline solution (4mg) via an identical spray device. Participants will be stratified for sex and then randomized to saline arm (The dose of saline will be (0.1 mL 0.9% sodium chloride intranasally), respectively. Investigators, staff, and participants will be blinded to the treatment options.
  Interventions: Behavioral: Active Virtual Reality; Behavioral: sham Virtual Reality; Other: No Intervention; Other: Saline
- Natural History (Other): Natural history group, where participants will not be given any drugs. Participants will be stratified for sex and then randomized to the Natural History group.
  Interventions: Behavioral: Active Virtual Reality; Behavioral: sham Virtual Reality; Other: No Intervention; Other: Natural history

INTERVENTIONS:
Behavioral: Active Virtual Reality — Participants will be assigned to an immersive VR environment.
  Other Names: Active VR
Behavioral: sham Virtual Reality — Participants will be assigned to a sham VR environment without the immersive experience.
  Other Names: Sham VR
Other: No Intervention — Participants will experience tonic pain tolerance tests without exposure to any environments.
Drug: Naloxone — 4mg of Naloxone will be administered (0.1 mL of 40 mg/ml naloxone solution given intranasally).
  A random allocation sequence will be independently generated by the UM Pharmacy. The Principal investigator will call for each experiment.
  Other Names: Naloxone Hydrochloride/Narcan Intranasal
  Arms: Naloxone
Other: Saline — Intranasal Normal Saline (0.1 mL 0.9% sodium chloride) will be administered shortly before beginning the fMRI experiment.
  A random allocation sequence will be independently generated by the UM Pharmacy. The Principal investigator will call for each experiment.
  Other Names: Placebo, Sodium chloride
  Arms: Saline
Other: Natural history — Participants will not be provided Naloxone or Saline.
  Arms: Natural History

SUMMARY:
This project examines, in chronic pain, the mechanisms of immersive virtual reality compared to the mechanisms of placebo hypoalgesia. The potential of developing new non-pharmacological premises for low-risk interventions for pain management is high.

DETAILED DESCRIPTION:
Virtual reality (VR) has been seen as an intervention for alleviating clinical chronic (and acute) pain. An approach to pain management utilizing VR presents opportunities for reducing pain and suffering by using immersive, aesthetic, and multisensory stimulation. Investigator will analyze the behavioral and neural mechanisms of active VR against sham VR as two methods that investigate descending pain modulation. Thus, the central hypothesis is that those who respond to placebos will likely respond to active VR. If VR-induced analgesia depends upon the release of endogenous opioids.

In this project, the investigators will determine the effects of VR at the neural and clinical levels directly for TMD participants, inviting participants from an existing Colloca Lab-based cohort phenotyped for diagnosis, grade, and low/high impact pain profiles and prospective TMD participants in collaboration with Johns Hopkins University. These participants have agreed to be recontacted for further research. Investigator will determine the role of the opioid tone (AIM1). In Aim 1, the investigators will determine the role of the endogenous opioid tone for VR-induced hypoalgesia in TMD participants using VR, tonic painful stimuli, and naloxone given intranasally with established mu-opioid receptor occupancy to determine how the opioid tone shapes VR-induced hypoalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-88 years)
* English speaker (written and spoken)
* Temporal Mandibular Disorder (TMD) for at least 3 months

Exclusion Criteria:

* Present or past degenerative neuromuscular disease
* Cardiovascular, neurological diseases, pulmonary abnormalities, kidney disease, liver disease, history of cancer within past 3 years
* Cervical pain other than TMD related (e.g. stenosis, radiculopathy)
* Any personal (or family first degree) history of mania, schizophrenia, or other psychoses
* Severe psychiatric condition (e.g., schizophrenia, bipolar disorders, autism) leading to hospitalization within the last 3 years.
* Use of antidepressants, ADHD medication, non-over-the-counter painkillers, methadone, benzodiazepines, barbiturates, and/or narcotics during the past 3 months
* Lifetime alcohol/drug dependence or alcohol/drug abuse in the past 3 months
* Pregnancy or breastfeeding
* Color-blindness
* Pain in jaw or temple in last 3 months due to toothache or infection
* Any facial trauma that has occurred in the last 6 weeks
* History of severe facial trauma in the last 3 months
* Impaired or uncorrected hearing
* Conditions that would interfere with the VR mask placement (e.g. trauma, burn, infection)
* Known history of severe motion sickness
* High blood pressure or symptomatic low blood pressure
* History of fainting
* History of angioedema
* Failed drug test (testing for opiates, cocaine, methamphetamines, amphetamines, and THC)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Ischemic pain endurance | one session lasting from 2 to 3 hours
  Increments in experimental ischemic pain endurance will be assessed using a timer (minutes of tolerance)

SECONDARY OUTCOMES:
Ischemic pain rating | one session lasting from 2 to 3 hours
  Increments in experimental ischemic pain endurance will be assessed using Visual Analogue Scale (VAS) (self-reported numbers) anchored from 0=no pain to 100=maximum tolerable pain. The VAS will be used every 10 seconds during the ischemic pain endurance task

CONTACTS AND LOCATIONS:
Overall Officials: Luana Colloca, MD/PhD/MS, Principal Investigator — University of Maryland Baltimore School of Nursing
Locations (1):
- Luana Colloca, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is neither intent nor plan to share IPD.

REFERENCES:
- [Background] Honzel E, Murthi S, Brawn-Cinani B, Colloca G, Kier C, Varshney A, Colloca L. Virtual reality, music, and pain: developing the premise for an interdisciplinary approach to pain management. Pain. 2019 Sep;160(9):1909-1919. doi: 10.1097/j.pain.0000000000001539. No abstract available. PMID 30817437
- [Background] Colloca L, Raghuraman N, Wang Y, Akintola T, Brawn-Cinani B, Colloca G, Kier C, Varshney A, Murthi S. Virtual reality: physiological and behavioral mechanisms to increase individual pain tolerance limits. Pain. 2020 Sep 1;161(9):2010-2021. doi: 10.1097/j.pain.0000000000001900. PMID 32345915
- [Background] Colloca L. The Placebo Effect in Pain Therapies. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:191-211. doi: 10.1146/annurev-pharmtox-010818-021542. Epub 2018 Sep 14. PMID 30216744
- [Background] Amanzio M, Benedetti F. Neuropharmacological dissection of placebo analgesia: expectation-activated opioid systems versus conditioning-activated specific subsystems. J Neurosci. 1999 Jan 1;19(1):484-94. doi: 10.1523/JNEUROSCI.19-01-00484.1999. PMID 9870976